CLINICAL TRIAL: NCT03225807
Title: Implementation of Lung Protective Ventilation in Patients With Acute Respiratory Failure
Acronym: IMPROVENT
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Colin Grissom, Principal Investigator, Intermountain Health Care, Inc.
Other Study IDs: 1050159
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Acute Respiratory Distress Syndrome; ARDS; Respiratory Distress Syndrome, Acute; Respiratory Insufficiency; Respiratory Distress Syndrome; Shock Lung; Severe Acute Respiratory Syndrome
Keywords: Intubated; Intubation; Ventilator; Ventilator-free days; Ventilator free days; Mechanical Ventilation; Meta-Analysis; Tidal Volume; Tidal Volumes; inflammation; cytokines; Pulmonary Infiltrate; Pulmonary Infiltrates; Low Tidal Volumes; Protective Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Severe Acute Respiratory Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a quality improvement study with the purpose of observing and measuring the effects of implementation of a proven standardized lung protective ventilation protocol in the new electronic medical record system iCentra across all Intermountain Healthcare hospitals. Approximately 14,000 records will be accessed for this study from a database of mechanically ventilated patients established for quality improvement purposes.

The investigators hypothesize that implementation of a standardized computerized lung protective ventilation protocol across all Intermountain Healthcare hospitals will be feasible, will decrease initial tidal volumes to the target 6 ml/kg PBW, and will improve outcomes.

The objectives of this study are to:

* Determine if the implementation of lung protective ventilation (with a 6 ml/kg PBW tidal volume ventilation protocol on initiation of mechanical ventilation) improves outcomes in patients with acute respiratory failure requiring mechanical ventilation
* Determine if the implementation of lung protective ventilation (with a 6 ml/kg PBW tidal volume ventilation protocol on initiation of mechanical ventilation) improves outcomes in the sub-group of patients with the acute respiratory distress syndrome (ARDS)
* Measure compliance with the implementation of a computerized lung protective ventilation protocol at 12 Intermountain Healthcare hospitals

DETAILED DESCRIPTION:
Study Design:

This is an observational quality improvement study comparing outcomes before, and after, implementation of a proven lung protective ventilation protocol in an electronic medical record system, iCentra, that will be implemented in phases across Intermountain Healthcare hospitals. A phased implementation with a two-month washout period will be used to evaluate the primary outcome of interest, ventilator free days (VFDs) to 28 days. Secondary outcomes will include: use of the protocol by clinicians, compliance with protocol instructions, hospital discharge disposition, hospital, 30-day, and 90-day mortality, time to first ICU activity, hospital length of stay, ICU length of stay, heath care utilization, quality of life, and costs of care. As the iCentra electronic medical record is implemented at Intermountain Healthcare hospitals, clinicians will have the opportunity to use the computerized lung protective ventilation protocol, or to order mechanical ventilation settings independently. This is an observational study designed to measure how often the computerized lung protective ventilation protocol will be ordered, compliance with the instructions of the protocol, and clinical outcomes among patients who are managed with the protocol. Physicians may choose to use the protocol on intubated patients requiring mechanical ventilation or they may choose to order other specific mechanical ventilator settings.

ELIGIBILITY:
Inclusion Criteria

1. Initiation of mechanical ventilation in the emergency department or intensive care unit at an Intermountain Healthcare hospital
2. Age ≥ 18 years

Exclusion Criteria

1. Transition to comfort care in the emergency department or on the same day of admission to the ICU
2. Death on the same day of admission to the emergency department or ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Selection Those to be enrolled must have respiratory failure requiring intubation and initiation of mechanical ventilation. Patients will be divided into two different groups: those patients who are managed with the computerized lung protective ventilation protocol as ordered by the attending physician and those patients managed with physician specified mechanical ventilation settings.
Sampling Method: Probability Sample
Enrollment: 8692 (Actual)
Dates: Start 2016-03; Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Ventilator free days to day 28 | 28 days

SECONDARY OUTCOMES:
30 day mortality | 30 days
90 day mortality | 90 days
Hospital discharge disposition | 30 days
Hospital mortality | 1 week
Time to first ICU activity | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Colin Grissom, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Colin Grissom, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared.

REFERENCES:
- [Derived] Grissom CK, Lanspa MJ, Groat D, Jacobs JR, Carpenter L, Kuttler KG, Leither L, Peltan ID, Brown SM, Srivastava R. Implementation of Lung-Protective Ventilation in Patients With Acute Respiratory Failure. Crit Care Med. 2023 Jun 1;51(6):797-807. doi: 10.1097/CCM.0000000000005840. Epub 2023 Mar 29. PMID 36988337

DOCUMENTS (1):
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03225807/Prot_000.pdf